CLINICAL TRIAL: NCT04275479
Title: Endocrine Diabetes Screening in Patients With Shwachman-Diamond Syndrome DIABETES/ ENDOCRINE SURVEILLANCE IN SDS
Brief Title: Diabetes/ Endocrine Surveillance in SDS
Status: Terminated | Type: Observational
Why Stopped: funding stopped
Sponsor: Washington University School of Medicine (Other)
Collaborators: Shwachman Diamond Syndrome Foundation (Unknown); Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201909102
Record Dates: First submitted 2020-02-10; First posted 2020-02-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Shwachman-Diamond Syndrome
Keywords: Shwachman-Diamond Syndrome; Atypical Diabetes; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Shwachman-Diamond Syndrome; Exocrine Pancreatic Insufficiency | interventions — Glucose Tolerance Test; Diet Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- SDS - without Diabetes diagnosis: SDS - without Diabetes diagnosis
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Other: Modified Oral Glucose Tolerance Test; Other: Modified Mixed Meal Tolerance Test; Device: Continuous Glucose Monitor; Other: Food Diary; Other: Medical History Questionnaires
- SDS with Diabetes Diagnosis: SDS with Diabetes Diagnosis
  Interventions: Other: Modified Mixed Meal Tolerance Test; Device: Continuous Glucose Monitor; Other: Food Diary; Other: Medical History Questionnaires
- Cystic Fibrosis (CF) patients data & lab results: De-identified data from age matched population norms, CF patients associated pancreatic insufficiency known or treated diabetes

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — This is a two step process. Subjects will be asked to fast overnight,(no food and only water to drink for at least 8 hours). Then when subjects arrive for the visit,participants will have blood drawn and be asked to drink a sugary liquid. One hour later, another blood sample will be drawn and after two hours a final blood sample will be drawn.
  Other Names: OGTT
  Groups: SDS - without Diabetes diagnosis
Other: Modified Oral Glucose Tolerance Test — The participant will be asked to fast overnight (no food and only water to drink for at least 8 hours). There will be no blood drawn during this test, participant will be asked to drink a sugary liquid and to remaining fasting (water only) for the two hour after finishing the drink.
  Other Names: Modified OGTT
  Groups: SDS - without Diabetes diagnosis
Other: Modified Mixed Meal Tolerance Test — The participant will be asked to fast overnight (no food and only water to drink for at least 8 hours). The participant will be given a meal supplement to drink in place of breakfast, for example Boost Plus. The participant will be asked to drink the meal supplement and to remaining fasting (water only) for the next two hours.
  Other Names: MMTT
  Groups: SDS - without Diabetes diagnosis; SDS with Diabetes Diagnosis
Device: Continuous Glucose Monitor — The participant will be provided a CGM device to wear for 10 days during the study period. The CGM will be blinded (meaning that the participant will not be able to see the results).
  Other Names: CGM
  Groups: SDS - without Diabetes diagnosis; SDS with Diabetes Diagnosis
Other: Food Diary — The participant will be asked to maintain a detailed food diary for 3 days during the 10 day study period.
  Groups: SDS - without Diabetes diagnosis; SDS with Diabetes Diagnosis
Other: Medical History Questionnaires — The participant will be asked to provide detailed medical history
  Groups: SDS - without Diabetes diagnosis; SDS with Diabetes Diagnosis

SUMMARY:
Shwachman-Diamond syndrome(SDS) is a rare autosomal recessive disorder involving primarily the Shwachman-Bodian-Diamond syndrome gene located on chromosome 7q11. The gene effects function of the 60S ribosome by interfering with the function of the Guanasine triphosphatase elongation factor 1 in the release of eukaryotic initiation factor 6 from the 60 S ribosomal subunit for translation initiation. Seventy five percent of the individual affected by the syndrome have a biallelic mutation (258+2T>C and 183-184T > CT). The syndrome results in defects primarily in the pancreas and bone marrow resulting in pancreatic insufficiency, leukopenia with an increased risk of infection and an increased risk for acute myelocytic leukemia. Animal models that have knocked out the function of the SBDS gene in the pancreas reveals at the pancreas at birth as well as the insulin producing cells in the pancreas are normal but subsequently developed fatty infiltration and apoptosis without inflammation resulting in pancreatic exocrine insufficiency with initially normal endocrine pancreatic function. The endocrine pancreatic function declines over time such that by 12 months of age these mice show a phenotype of impaired glucose tolerance. The finding of early onset diabetes is not yet considered a manifestation of this genetic defect but likely is occurring. This study is designed to assist in understanding the prevalence of glucose abnormalities in this syndrome.

Exocrine pancreatic insufficiency leading to diabetes is a common hallmark of cystic fibrosis and cystic fibrosis related diabetes. Prevalence of glucose abnormalities in diabetes is a approaching 50% by the 2nd and 3rd decade of life in this disorder. The cystic fibrosis Foundation recommend screening for diabetes utilizing an oral glucose tolerance by the age of 10. Early diagnosis of diabetes in the syndrome as resulted in improved outcomes for patients with cystic fibrosis. It is my expectation that the prevalence of diabetes will be similar in SBDS patients. A small study performed I had the University of Cincinnati showed glucose abnormalities to occur in 5/20 individuals with the classic mutation.

Investigators propose to screen patients with the classic mutation for diabetes and endocrine disease utilizing continuous glucose monitoring over a 14 day period in addition to baseline fasting blood tests for insulin, GAD 65 antibody, Fructosamine, A1c and C peptide.

DETAILED DESCRIPTION:
The purpose of the study is to learn about how common early onset diabetes and other endocrine issues occur in people who have been diagnosed with SDS.

Study procedures include:

For participants with SDS:

obtaining informed consent/assent; obtaining medical & medication history, including history of diabetes, review of medical records and lab results for confirmation of diagnosis and inclusion/exclusion assessment; performance of a standard oral glucose tolerance test (OGTT) to be performed at a center close to the participants home, a modified oral glucose tolerance test and a modified mixed meal tolerance test to be performed by participant at home with phone access to study staff for directions, blood draws performed at a local lab or local physician office or other medical center in close proximity to the participants home. Completion of on-line, or in the case of no computer access - paper, questionnaires completed by the participant/parent to collect medical and health history, parents/siblings will be asked to complete a health history, 3 day food diary completed by participant/parent; phone calls; wearing of blinded continuous glucose monitoring device for 14 days; medical records release, 3-day diet diary; Additional optional biological specimens to look at cell free DNA and future biomarkers of endoplasmic reticulum stress in the beta cells of the pancreas will be obtained and stored for future study Parent(s) and/or siblings if willing and consented, will complete on-line medical history questionnaire and provide medical record release.

Data to be obtained from on-going study for subjects with Cystic Fibrosis

ELIGIBILITY:
Inclusion Criteria:

Population 1: SDS and non-diabetic

* Age: 3 years of age and older to allow for baseline blood to be drawn. The Cystic Fibrosis group has seen glucose abnormalities well before age 10 but recommends screening after age 10. Investigators are attempting to define the population and will screen starting at age 3 to get a baseline data set.
* Willing to provide consent/ assent
* Stable health in the last month- i.e. not hospitalized/ ill in the last 6 weeks
* Patients should have been on stable medications for at least 4 weeks prior to testing - This includes neupogen and other white cell stimulators.
* Classic SBDS mutation with pancreatic insufficiency as determined by medical history.
* Able/willing to have a standard OGTT and modified OGTT
* Able/ willing to wear a Libre- Pro sensor and have sensor returned. If not willing to wear CGM- willing to do a standard OGTT as described.
* Not currently on diabetic therapy or labeled as diabetic.
* Willing to complete a health survey in regard to the SBDS and endocrine History

Population 2: SDS and Labeled as diabetic

* Age greater than 3
* If labeled as diabetic - obtain data for age of onset and treatment utilized for the diabetes
* Willing to provide consent/ assent and complete health survey for SBDS and endocrine history
* Willing/able to wear 14 day blinded Libre-Pro to assess the response to current therapy and food diary.
* Willing to provide Fasting labs as outlined above for the group- no OGT, just the mixed meal tolerance test

Population 1 and 2 Future Sub-study: Assess alpha cell and insulin dynamic response

* Participant in primary study who agree to the sub-study
* Willing to travel to St. Louis for clamp procedure.
* Budget will determine the actual number to be screened.
* Travel will be included.

Population 3: Control groups

* Other control groups for the study will be age matched population norms, Cystic Fibrosis patients associated pancreatic insufficiency known or treated diabetes.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample, SDS Registry
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Systematically assess the prevalence of diabetes or glucose intolerance in participants with the classic biallelic mutation | 1 Year
  Aim 1
Longitudinal screening of the enrolled population to assess the prevalence of diabetes or glucose intolerance | Through study completion, an average of 3 years
  Aim 2
Assess individuals who have previously been diagnosed with diabetes in regard to age of onset, complications and the treatments utilized. | 1 year
  Aim 3
Assist families and patients in understanding their diet and fine tuning their approach to carbohydrates and fat in the diet | 1 year
  Aim 4
Share data with the current SBDS Registry | Through study completion, and average of 3 years
  Aim 5

CONTACTS AND LOCATIONS:
Overall Officials: Garry Tobin, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finch AJ, Hilcenko C, Basse N, Drynan LF, Goyenechea B, Menne TF, Gonzalez Fernandez A, Simpson P, D'Santos CS, Arends MJ, Donadieu J, Bellanne-Chantelot C, Costanzo M, Boone C, McKenzie AN, Freund SM, Warren AJ. Uncoupling of GTP hydrolysis from eIF6 release on the ribosome causes Shwachman-Diamond syndrome. Genes Dev. 2011 May 1;25(9):917-29. doi: 10.1101/gad.623011. PMID 21536732
- [Background] Menne TF, Goyenechea B, Sanchez-Puig N, Wong CC, Tonkin LM, Ancliff PJ, Brost RL, Costanzo M, Boone C, Warren AJ. The Shwachman-Bodian-Diamond syndrome protein mediates translational activation of ribosomes in yeast. Nat Genet. 2007 Apr;39(4):486-95. doi: 10.1038/ng1994. Epub 2007 Mar 11. PMID 17353896
- [Background] Tourlakis ME, Zhong J, Gandhi R, Zhang S, Chen L, Durie PR, Rommens JM. Deficiency of Sbds in the mouse pancreas leads to features of Shwachman-Diamond syndrome, with loss of zymogen granules. Gastroenterology. 2012 Aug;143(2):481-92. doi: 10.1053/j.gastro.2012.04.012. Epub 2012 Apr 14. PMID 22510201
- [Background] Moran A, Brunzell C, Cohen RC, Katz M, Marshall BC, Onady G, Robinson KA, Sabadosa KA, Stecenko A, Slovis B; CFRD Guidelines Committee. Clinical care guidelines for cystic fibrosis-related diabetes: a position statement of the American Diabetes Association and a clinical practice guideline of the Cystic Fibrosis Foundation, endorsed by the Pediatric Endocrine Society. Diabetes Care. 2010 Dec;33(12):2697-708. doi: 10.2337/dc10-1768. No abstract available. PMID 21115772
- [Background] Dror Y, Donadieu J, Koglmeier J, Dodge J, Toiviainen-Salo S, Makitie O, Kerr E, Zeidler C, Shimamura A, Shah N, Cipolli M, Kuijpers T, Durie P, Rommens J, Siderius L, Liu JM. Draft consensus guidelines for diagnosis and treatment of Shwachman-Diamond syndrome. Ann N Y Acad Sci. 2011 Dec;1242:40-55. doi: 10.1111/j.1749-6632.2011.06349.x. PMID 22191555
- [Background] Myers KC, Rose SR, Rutter MM, Mehta PA, Khoury JC, Cole T, Harris RE. Endocrine evaluation of children with and without Shwachman-Bodian-Diamond syndrome gene mutations and Shwachman-Diamond syndrome. J Pediatr. 2013 Jun;162(6):1235-40, 1240.e1. doi: 10.1016/j.jpeds.2012.11.062. Epub 2013 Jan 8. PMID 23305959
- [Background] Diabetes Care. Introduction. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S1-2. doi: 10.2337/dc10-S001. No abstract available. PMID 20042770
- [Background] Jivani N, Torrado-Jule C, Vaiselbuh S, Romanos-Sirakis E. A unique case of Shwachman-Diamond syndrome presenting with congenital hypopituitarism. J Pediatr Endocrinol Metab. 2016 Nov 1;29(11):1325-1327. doi: 10.1515/jpem-2016-0299. PMID 27754968
- [Background] Gana S, Sainati L, Frau MR, Monciotti C, Poli F, Cannioto Z, Comelli M, Danesino C, Minelli A. Shwachman-Diamond syndrome and type 1 diabetes mellitus: more than a chance association? Exp Clin Endocrinol Diabetes. 2011 Nov;119(10):610-2. doi: 10.1055/s-0031-1275699. Epub 2011 May 6. PMID 21553366
- [Background] Akdogan MF, Altay M, Denizli N, Gucun M, Tanrikulu S, Duranay M. A rare case: Shwachman-Diamond syndrome presenting with diabetic ketoacidosis. Endocrine. 2011 Aug;40(1):146-7. doi: 10.1007/s12020-011-9460-7. No abstract available. PMID 21448781
- [Background] Besser RE, Shields BM, Casas R, Hattersley AT, Ludvigsson J. Lessons from the mixed-meal tolerance test: use of 90-minute and fasting C-peptide in pediatric diabetes. Diabetes Care. 2013 Feb;36(2):195-201. doi: 10.2337/dc12-0836. Epub 2012 Oct 30. PMID 23111058
- [Background] Al Hayek AA, Robert AA, Al Dawish MA. Evaluation of FreeStyle Libre Flash Glucose Monitoring System on Glycemic Control, Health-Related Quality of Life, and Fear of Hypoglycemia in Patients with Type 1 Diabetes. Clin Med Insights Endocrinol Diabetes. 2017 Dec 10;10:1179551417746957. doi: 10.1177/1179551417746957. eCollection 2017. PMID 29270042
- [Background] Boudreau V, Lehoux Dubois C, Desjardins K, Mailhot M, Tremblay F, Rabasa-Lhoret R. Sensitivity and specificity of cystic fibrosis-related diabetes screening methods: which test should be the reference method? J Pediatr Endocrinol Metab. 2017 Aug 28;30(8):885-887. doi: 10.1515/jpem-2017-0122. No abstract available. PMID 28742521
- [Background] Brugha R, Wright M, Nolan S, Bridges N, Carr SB. Quantifying fluctuation in glucose levels to identify early changes in glucose homeostasis in cystic fibrosis. J Cyst Fibros. 2018 Nov;17(6):791-797. doi: 10.1016/j.jcf.2017.12.004. Epub 2018 Jan 10. PMID 29329721
- [Background] Clemente Leon M, Bilbao Gasso L, Moreno-Galdo A, Campos Martorrell A, Gartner Tizzano S, Yeste Fernandez D, Carrascosa Lezcano A. Oral glucose tolerance test and continuous glucose monitoring to assess diabetes development in cystic fibrosis patients. Endocrinol Diabetes Nutr (Engl Ed). 2018 Jan;65(1):45-51. doi: 10.1016/j.endinu.2017.08.008. Epub 2017 Nov 12. English, Spanish. PMID 29137964
- [Background] Deja G, Kleczek M, Chumiecki M, Strzala-Kleczek A, Deja R, Jarosz-Chobot P. The usefulness of the FlashStyle Libre system in glycemic control in children with type 1 diabetes during summer camp. Pediatr Endocrinol Diabetes Metab. 2018;24(1):11-19. doi: 10.18544/PEDM-24.01.0098. PMID 30083658
- [Background] Giani E, Macedoni M, Barilli A, Petitti A, Mameli C, Bosetti A, Cristiano A, Radovanovic D, Santus P, Zuccotti GV. Performance of the Flash Glucose Monitoring System during exercise in youth with Type 1 diabetes. Diabetes Res Clin Pract. 2018 Dec;146:321-329. doi: 10.1016/j.diabres.2018.10.001. Epub 2018 Oct 9. PMID 30312715
- [Background] Hoss U, Budiman ES. Factory-Calibrated Continuous Glucose Sensors: The Science Behind the Technology. Diabetes Technol Ther. 2017 May;19(S2):S44-S50. doi: 10.1089/dia.2017.0025. PMID 28541139
- [Background] Landau Z, Abiri S, Gruber N, Levy-Shraga Y, Brener A, Lebenthal Y, Barash G, Pinhas-Hamiel O, Rachmiel M. Use of flash glucose-sensing technology (FreeStyle Libre) in youth with type 1 diabetes: AWeSoMe study group real-life observational experience. Acta Diabetol. 2018 Dec;55(12):1303-1310. doi: 10.1007/s00592-018-1218-8. Epub 2018 Aug 31. PMID 30171412
- [Background] Massa GG, Gys I, Op 't Eyndt A, Bevilacqua E, Wijnands A, Declercq P, Zeevaert R. Evaluation of the FreeStyle(R) Libre Flash Glucose Monitoring System in Children and Adolescents with Type 1 Diabetes. Horm Res Paediatr. 2018;89(3):189-199. doi: 10.1159/000487361. Epub 2018 Mar 27. PMID 29587254
- [Background] Edge J, Acerini C, Campbell F, Hamilton-Shield J, Moudiotis C, Rahman S, Randell T, Smith A, Trevelyan N. An alternative sensor-based method for glucose monitoring in children and young people with diabetes. Arch Dis Child. 2017 Jun;102(6):543-549. doi: 10.1136/archdischild-2016-311530. Epub 2017 Jan 30. PMID 28137708
- See also: Shwachman-Diamond Syndrome Foundation — https://shwachman-diamond.org/
- See also: Washington University Research Participant Registry — https://sites.wustl.edu/wuvfh/
- See also: Washington University- Understanding Clinical Trials — https://wuphysicians.wustl.edu/clinical-trials/understanding-clinical-trials